CLINICAL TRIAL: NCT00596687
Title: RAndomized Study of Basal Bolus Insulin Therapy in the Inpatient Management of Patients With Type 2 Diabetes Undergoing General Surgery (RABBIT 2 Surgery)
Brief Title: Basal Bolus Insulin Versus SSRI in Type 2 Diabetes Undergoing General Surgery
Acronym: RABBIT 2-SX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005062; e5062
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes; Inpatient Hyperglycemia
Keywords: diabetes; post-op complications; inpatient hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine; Insulin; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Glargine once daily plus glulisine given before meals plus supplemental glulisine for BG > 140
  Interventions: Drug: Insulin glargine; Drug: Insulin glulisine
- 2 (Active Comparator): Sliding scale regular insulin four-times daily achs.
  Interventions: Drug: Regular insulin

INTERVENTIONS:
Drug: Insulin glargine — Insulin glargine once daily SQ
  Other Names: Lantus
  Arms: 1
Drug: Regular insulin — Sliding scale regular insulin SQ four-times daily before meals or every 6 hours if patient NPO
  Other Names: Novolin R
  Arms: 2
Drug: Insulin glulisine — scheduled glulisine given SQ at mealtime TID; none given if patient NPO
  Other Names: Apidra
  Arms: 1

SUMMARY:
High blood glucose levels in surgical patients with diabetes are associated with increased risk of medical complications and death. Improved glucose control with insulin injections may improve clinical outcome and prevent some of the hospital complications. In patients who have undergone surgery, high blood glucose increases the risk of wound infection, kidney failure and death. It is not known; however, what is the best insulin regimen in patients who will undergo surgery. The use of repeated injections of regular insulin is commonly used for glucose control in hospitalized patients with diabetes. Recently, the combination of Lantus® and Apidra® insulins has been shown to improve glucose control with lower rate of hypoglycemia (low blood sugar). We hypothesize that in patients with type 2 diabetes admitted to general surgery wards, treatment with once daily glargine (Lantus) plus supplemental glulisine insulin (Apidra®) will produce better glycemic control and a lower rate of hospital complications than treatment with regular insulin per sliding scale (SSRI). The present study aims to determine which insulin treatment is best for glucose control in hospitalized patients with diabetes. Glargine and glulisine insulins are approved for use in the treatment of patients with diabetes by the FDA.

Subjects included in the study will have type 2 diabetes and be admitted to Grady Memorial Hospital, Veterans Administration Medical Center, and Emory University Hospital, Atlanta, Georgia. A total of ~94 patients will be recruited at each institution.

A post-hoc cost analysis of hospitalization costs and charges of the Rabbit surgery trial will be completed in order to determine differences in hospitalization cost between basal bolus insulin and SSI regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years admitted to a general surgery service.
2. Patients admitted for non-cardiac elective or emergency surgery or trauma.
3. A known history of type 2 diabetes mellitus > 3 months, receiving either diet alone or any combination of oral antidiabetic agents (sulfonylureas, metformin, thiazolidinediones).
4. Subjects must have an admission blood glucose > 140 mg and < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 mEq/L or positive serum or urinary ketones).

Exclusion Criteria:

1. Subjects with increased blood glucose concentration, but without a known history of diabetes (stress hyperglycemia).
2. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria.
3. Acute critical illness or CABG surgery expected to require prolonged admission to a critical care unit (ICU, CCU, SICU, Neuro ICU).
4. Patients with clinically relevant hepatic disease or impaired renal function, as shown by a serum creatinine ≥ 3.5 mg/dl.
5. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
6. Female subjects are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Result] Umpierrez GE, Smiley D, Jacobs S, Peng L, Temponi A, Mulligan P, Umpierrez D, Newton C, Olson D, Rizzo M. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes undergoing general surgery (RABBIT 2 surgery). Diabetes Care. 2011 Feb;34(2):256-61. doi: 10.2337/dc10-1407. Epub 2011 Jan 12. PMID 21228246
- [Derived] Umpierrez GE, Jones S, Smiley D, Mulligan P, Keyler T, Temponi A, Semakula C, Umpierrez D, Peng L, Ceron M, Robalino G. Insulin analogs versus human insulin in the treatment of patients with diabetic ketoacidosis: a randomized controlled trial. Diabetes Care. 2009 Jul;32(7):1164-9. doi: 10.2337/dc09-0169. Epub 2009 Apr 14. PMID 19366972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled patients with a BG 140-400 mg/dL with DM for more than 3 months,aged 18-80 yo, treated with diet alone, any combination of oral antidiabetic agents, or lowdose insulin in 2008-2009. Study was conducted at Grady Memorial Hospital,Emory University Hospitaland the Veterans Administration Medical Center.
Pre-assignment Details: Exclusion criteria included hyperglycemia without a known history of diabetes, cardiac surgery, clinically relevant hepatic disease or impaired renal function (serum creatinine ≥3.0 mg/dL), history of diabetic ketoacidosis (20), pregnancy, and any mental condition rendering the subject unable to give informed consent.
Groups:
- Basal Bolus: Glargine and rapid-acting mealtime insulin plus supplemental glulisine. A total of 0.5 units of insulin/day given, half as basal glargine insulin once a day and the other half as mealtime glulisine given three times a day at meals.
- SSRI: Sliding scale regular insulin four-times daily if blood glucose > 140 before meals and at bedtime. The sliding scale regimen was per the hospital protocol.
Period: Overall Study
Arm/Group | Basal Bolus | SSRI
Started | 118 | 116
Completed | 104 | 107
Not Completed | 14 | 9
Not completed — < 24 hours of insulin treatment | 8 | 6
Not completed — continuous insulin infusion during TPN | 2 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — cancelled surgery | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Basal Bolus: Glargine and rapid-acting mealtime insulin plus supplemental glulisine
- SSRI: Sliding scale regular insulin four-times daily.
- Total: Total of all reporting groups
Arm/Group | Basal Bolus | SSRI | Total
Number analyzed (Participants) | 104 | 107 | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 101 | 102 | 203
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 57 (10) | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 54 | 104
  Male | 54 | 53 | 107
Region of Enrollment [Number; unit: participants]
  United States | 104 | 107 | 211

OUTCOME MEASURES:

1. Secondary Outcome: # Participants With Hypoglycemic Events
Description: number of participants in the treatment arms with of hypoglycemic events (< 70 mg/dl)
Time Frame: hospital stay days 2-10
Measure: Number; unit: participants
Arm/Group | Basal Bolus | SSRI
Number analyzed (Participants) | 104 | 107
participants | 24 | 5

2. Primary Outcome: Mean Blood Glucose Concentration
Description: blood glucose concentration in the intervention groups after second day of treatment to up to 10 days of treatment
Time Frame: hospital stay days 2-10
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Basal Bolus | SSRI
Number analyzed (Participants) | 104 | 107
mg/dl | 145 (32) | 172 (46)

ADVERSE EVENTS:
Time Frame: during hospital days 1-10
Arm/Group | Basal Bolus | SSRI
Serious Adverse Events (participants affected / at risk) | 24/104 | 5/107
Other Adverse Events (participants affected / at risk) | 0/104 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal Bolus (N=104) | SSRI (N=107)
Hypoglycemia < 70 mg/dl (Metabolism and nutrition disorders) | 24 (24) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No